CLINICAL TRIAL: NCT00797836
Title: Cost-effectiveness of Quantiferon Gold in VITRO Test of T-lymphocytic Response for Detection of Latent Tuberculosis in At-risk Healthcare Workers
Brief Title: Quantiferon for Detection of Latent Tuberculosis in Healthcare Workers
Acronym: QUANTIPS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: P070312; STIC AOM04013 (Other: French Ministry)
Record Dates: First submitted 2008-11-24; First posted 2008-11-25 (Estimated); Last update posted 2012-01-10 (Estimated); Status verified 2008-11

CONDITIONS: Tuberculosis
Keywords: Occupational Diseases; Tuberculosis; Tuberculin Test; Immunoassay
MeSH Terms: conditions — Tuberculosis; Occupational Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Quantiferon Gold (Experimental)
  Interventions: Procedure: Quantiferon Gold

INTERVENTIONS:
Procedure: Quantiferon Gold — Interferon-gama release assay evaluating tuberculosis-specific T-lymphocytic response
  Health Personnel Hospitals, General Occupational Diseases/*epidemiology/*statistics & numerical data Occupational Exposure/*statistics & numerical data
  Tuberculosis/*diagnosis/*epidemiology/prevention & control Immunologic Tests/methods/*standards Disease Transmission, Horizontal/*statistics & numerical data Patient Isolation
  Tuberculin Test/standards/*methods Immunoassay/methods/*standards T-Lymphocytes/immunology Interferon Type II/*blood/*analysis
  *Reagent Kits, Diagnostic
  Mass Screening/*methods Incidence Follow-Up Studies Comparative Study Sensitivity and Specificity Risk Assessment/*methods
  Other Names: Interferon-gama; evaluating tuberculosis-specific T-lymphocytic response

SUMMARY:
The accuracy of tuberculin skin test (TST) for detecting latent tuberculosis is limited in countries with a high proportion of population having received vaccination with the BCG. We aim to determine the cost-effectiveness of Quantiferon gold (QTFG), compared to BCG vaccine to detect latent tuberculosis in exposed healthcare workers (HCWs)

DETAILED DESCRIPTION:
The QUANTIPS study includes two components:

1. survey of HCWs working in high-risk units (respiratory diseases or infectious diseases with at least 5 case of smear-positive pulmonary tuberculosis par year) from 14 University hospitals in France
2. Follow-up of HCWs with unexpected exposure to a patient with contagious tuberculosis (delay in respiratory isolation of a smear-positive patient) in 4 University hospitals Main objective: Therapeutic impact of tuberculosis screening using TST compared to QFTG. The impact is defined by the decision to treat of not a HCW with latent tuberculosis using QFTG, compared to the decision which would have been based on TST alone

Secondary objectives:

* Cost-effectiveness of replacing TST by QFTG
* Prevalence and incidence of latent tuberculosis in exposed HCWs (Part 1)
* Incidence of latent tuberculosis in HCWs exposed to an index case (part 2) Inclusion: HCWs who volunteer to participate in units with at least 5 patients with smear-positive tuberculosis each year (Group 1), HCWs exposed to a smear-positive patient non isolated at hospital admission (Group 2) Study population: 2000 (Group 1) and 600 (Group 2) HCWs Study duration: inclusion during 3 months, follow-up of one year (Group 1 ); Inclusion for one year, with a 3-month follow up (Group 2)

Study exams:

* Group 1 : TST, QFTG, chest radiography at baseline and after one year
* Group 2 : TST, QFTG, chest radiography at baseline (within 3 weeks after exposure) and after 3 months

Endpoints:

* therapeutic decision regarding tuberculosis treatment, with a cost-effectiveness analysis (Markov's modelling)
* prevalence and incidence of latent tuberculosis

ELIGIBILITY:
INCLUSION CRITERIA:

Group 1:

* Healthcare worker volunteering for the study
* Stable (expected employment in the unit > one year)
* Working in a high-risk units for tuberculosis (at least 5 cases of smear-positive pulmonary tuberculosis per year)

Group 2 :

* Healthcare worker volunteering for the study
* With an unexpected exposure to a patient with contagious tuberculosis (delay in respiratory isolation of a smear-positive patient)

EXCLUSION CRITERIA:

* No informed consent
* Age < 18 years
* Employment in this unit < one year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1024 (Actual)
Dates: Start 2008-11; Primary Completion 2010-10 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Therapeutic impact of tuberculosis screening using QFTG compared to TST. The impact is defined by the decision to treat of not a HCW with latent tuberculosis using QFTG, compared to the decision which would have been based on TST alone | 18 months

SECONDARY OUTCOMES:
Cost-effectiveness of replacing TST by QFTG | 18 months
Prevalence and incidence of latent tuberculosis in exposed HCWs (Group 1) | 18 months
Incidence of latent tuberculosis in HCWs exposed to an index case (Group 2) | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Guislaine CARCELAIN, Dr, Study Chair — Assistance Publique - Hôpitaux de Paris
Locations (1):
- CHU Bichat Claude Bernard, Paris, Île-de-France Region, France

REFERENCES:
- [Derived] Lucet JC, Abiteboul D, Estellat C, Roy C, Chollet-Martin S, Tubach F, Carcelain G; QUANTIPS Study Group. Interferon-gamma release assay vs. tuberculin skin test for tuberculosis screening in exposed healthcare workers: a longitudinal multicenter comparative study. Infect Control Hosp Epidemiol. 2015 May;36(5):569-74. doi: 10.1017/ice.2015.19. Epub 2015 Feb 16. PMID 25682769